CLINICAL TRIAL: NCT03861962
Title: Re-evaluation of Donor-specific Anti-HLA Alloantibodies Immunoassay After Organ Transplantation, From Antigen Level to Epitope Level: a Track to Improve Organ Allocation
Brief Title: Re-evaluation of Donor-specific Anti-HLA Alloantibodies Immunoassay After Organ Transplantation, From Antigen Level to Epitope Level
Acronym: ACORG-HLA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI16035HLJ
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-02

CONDITIONS: Organ Transplantation
Keywords: serum-specific donor antibodies (DSA); human leukocyte antigens (HLA); organ allocation; epitope level

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: DNA sequencing called "new generation" (or NGS) — Redo HLA-typings with a method exploring all the genes (add DQA1, DRB3 / 4/5, DPB1 and DPA1), i.e. DNA sequencing called "new generation", when this has not been done after the graft as part of the standard care

SUMMARY:
Transplantation is the only treatment for end-stage organ dysfunction, with dialysis for the kidney. However, donor / recipient (D / R) tissue incompatibility accounts for the majority of long-term graft losses, through the development of serum-specific donor antibodies (DSA) to human leukocyte antigens (HLA) of donor, with a prevalence of about 10% at 2 years and 20% at 5 years.

DSA immunization is very often directed against one or a few of the donor's incompatible antigens, suggesting that epitopes (and antigens) are not all equally immunogenic. Identifying HLA epitopes that cause the most and the least immunization would help refine the graft distribution to better manage a limited resource by defining the D / R combinations to avoid or promote. Since the immunogenicity of an HLA epitope depends on the HLA of the recipient given the properties of the epitopes mentioned above, a very large cohort is needed to understand this question. To do so, it is necessary to redo these typings with a method exploring all the genes (add DQA1, DRB3 / 4/5, DPB1 and DPA1) when this has not been done after the graft as part of the standard care. This has become possible since 3 years by DNA sequencing called "new generation" (or NGS), a method that is supplanting all others for the medical care of patients in transplantation.

This study is a retrospective cohort study with 5-year follow-up. The investigators' main objective is to evaluate the predictive value of the number of mismatched HLA epitopes for the development of DSA anti-HLA de novo at 2 years. The investigators' secondary objectives are to evaluate this parameter at 5 and 8 years to determine which epitope mismatches should be favored / avoided in the future.

ELIGIBILITY:
Inclusion Criteria:

* patients (adults and children)
* patients recipients in France from 2008 to 2015 of a first kidney transplant / heart / lung / liver donor living or deceased, non-immunized anti-HLA before the transplant
* patients having preserved their graft > 2 years
* having agreed to the use for research purposes in transplantation of the remains of the DNA and serum samples taken as part of the care of which the remains are available

Exclusion Criteria:

* no inclusion if one of the inclusion criteria is not met

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (adults and children) récipients of a first kidney transplant / heart / lung / liver donor living or deceased,non-immunized anti-HLA before the transplant, having preserved their graft > 2 years will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of serum-specific donor antibodies (DSA) | at 2 years after organ transplantation
  Proportion of serum-specific donor antibodies (DSA) regarding epitope mismatches

SECONDARY OUTCOMES:
Proportion of dnDSA anti-HLA | at 2 years after organ transplantation
Proportion of dnDSA anti-HLA | at 5 years after organ transplantation
Proportion of dnDSA anti-HLA | at 8 years after organ transplantation
Proportion of non-DSA anti-HLA antibodies | at 2 years after organ transplantation
Proportion of non-DSA anti-HLA antibodies | at 5 years after organ transplantation
Proportion of non-DSA anti-HLA antibodies | at 8 years after organ transplantation
Proportion of both total and HLA class I or class II dnDSA by HLA locus (A, B, C, DRB1, DRB3 / 4/5, DQB1, DQA1, DPB1, DPA1) , by HLA antigen, by epitope, for all types of organs and by organ type | at 2 years after organ transplantation
Proportion of both total and HLA class I or class II dnDSA by HLA locus (A, B, C, DRB1, DRB3 / 4/5, DQB1, DQA1, DPB1, DPA1) , by HLA antigen, by epitope, for all types of organs and by organ type | at 5 years after organ transplantation
Proportion of both total and HLA class I or class II dnDSA by HLA locus (A, B, C, DRB1, DRB3 / 4/5, DQB1, DQA1, DPB1, DPA1) , by HLA antigen, by epitope, for all types of organs and by organ type | at 8 years after organ transplantation
Number of dnDSA anti-HLA both total and by HLA class (class I versus class II), by HLA locus (A, B, C, DRB1, DRB3 / 4/5, DQB1, DQA1, DPB1, DPA1), by HLA antigen, for all organ types and organ type | at 2 years after organ transplantation
Number of dnDSA anti-HLA both total and by HLA class (class I versus class II), by HLA locus (A, B, C, DRB1, DRB3 / 4/5, DQB1, DQA1, DPB1, DPA1), by HLA antigen, for all organ types and organ type | at 5 years after organ transplantation
Number of dnDSA anti-HLA both total and by HLA class (class I versus class II), by HLA locus (A, B, C, DRB1, DRB3 / 4/5, DQB1, DQA1, DPB1, DPA1), by HLA antigen, for all organ types and organ type | at 8 years after organ transplantation
Distribution of anti-HLA dnDSA by targeted epitope and antigen (to define immunodominant and non-immunodominant epitopes and antigens), both total and by HLA class (class I versus class II), by HLA locus for all types of organs and organ type | at 2 years after organ transplantation
Distribution of anti-HLA dnDSA by targeted epitope and antigen (to define immunodominant and non-immunodominant epitopes and antigens), both total and by HLA class (class I versus class II), by HLA locus for all types of organs and organ type | at 5 years after organ transplantation
Distribution of anti-HLA dnDSA by targeted epitope and antigen (to define immunodominant and non-immunodominant epitopes and antigens), both total and by HLA class (class I versus class II), by HLA locus for all types of organs and organ type | at 8 years after organ transplantation
Distribution of strength anti-HLA dnDSA measured by mean fluorescence intensity to identify the immunodominant DSA, both global and by class, by HLA locus by HLA antigen, by epitope, for all types of organs and organ type | at 2 years after organ transplantation
Distribution of strength anti-HLA dnDSA measured by mean fluorescence intensity to identify the immunodominant DSA, both global and by class, by HLA locus by HLA antigen, by epitope, for all types of organs and organ type | at 5 years after organ transplantation
Distribution of strength anti-HLA dnDSA measured by mean fluorescence intensity to identify the immunodominant DSA, both global and by class, by HLA locus by HLA antigen, by epitope, for all types of organs and organ type | at 8 years after organ transplantation
Strength in mean fluorescence intensity of dnDSA anti-HLA de novo specific epitopes of epitopes DQbeta, DQalpha and composites (DQbeta + DQalpha) by antigen DQ | at 2 years after organ transplantation
Strength in mean fluorescence intensity of dnDSA anti-HLA de novo specific epitopes of epitopes DQbeta, DQalpha and composites (DQbeta + DQalpha) by antigen DQ | at 5 years after organ transplantation
Strength in mean fluorescence intensity of dnDSA anti-HLA de novo specific epitopes of epitopes DQbeta, DQalpha and composites (DQbeta + DQalpha) by antigen DQ | at 8 years after organ transplantation
Survival of the graft | at 5 years after organ transplantation
Survival of the graft | at 8 years after organ transplantation
Overall survival | at 5 years after organ transplantation
Overall survival | at 8 years after organ transplantation

IPD SHARING:
Plan to Share IPD: Undecided